CLINICAL TRIAL: NCT06230406
Title: Role of T-Mem GEne in the Molecular Pathogenesis of Atherosclerosis
Brief Title: T-Mem GEne in Atherosclerosis
Acronym: GEMMA
Status: Recruiting | Type: Observational
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Daniela Mazzaccaro, Vascular Surgeon, Researcher, PI, IRCCS Policlinico S. Donato
Other Study IDs: GEMMA V1 - 35/int/2023
Record Dates: First submitted 2023-12-27; First posted 2024-01-30 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Vascular tissue, blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: surgery for artherial and/or venous diseases — collection of vascular samples from surgery and blood samples

SUMMARY:
Atherosclerosis is the main cause of cardiovascular diseases and is characterized by the progressive accumulation of lipids and inflammatory cells such as macrophages and lymphocytes within the vessel wall of large and medium-sized arteries, forming the so-called "atherosclerotic plaques". The formation process of these lesions is different depending on the age, genetics and physiological state of the individual affected. Furthermore, behavioral factors and the lifestyle of each individual play a key role, which can lead to the presence of a series of pro-atherosclerotic pathologies and risk factors, such as in particular systemic arterial hypertension, dyslipidemia, hyperglycemia and cigarette smoking. However, the precise molecular mechanisms underlying this pathogenetic process are still under investigation.

The results of a study conducted in the past in collaboration between the U.O. have recently been published. of Vascular Surgery and the laboratory of Dr. I. Zucchi of the Institute of Biomedical Technologies of the CNR of Milan Segrate (Protocol GEMMA NUOVA, 16/int/2016), which describes that the overexpression of a newly identified gene (TMEM230) it may have a role in the formation of atherosclerotic vascular disorders, but it is still unclear how the expression of this gene is modulated in vivo.

Knowledge of these factors would increase the knowledge of the molecular mechanisms underlying atherosclerosis and could represent a possible target for prevention and targeted pharmacological treatment, with consequent potential reduction in disability or mortality from cardiovascular diseases.

DETAILED DESCRIPTION:
The proposed study aims to analyze, in patients suffering from vascular pathologies, the modulation of the expression of the TMEM230 gene, identified in the laboratory of Dr. I. Zucchi of the Institute of Biomedical Technologies (CNR of Milan Segrate), and its role in the molecular mechanisms of atherosclerosis.

This collaboration aims to collect a series of patients with different vascular pathologies.

This is a transversal genetic study, which involves the analysis of approximately 12 samples of vascular tissue of various types coming from the intraoperative removal of material that is normally disposed of in appropriate containers for biological waste. In particular, the vascular samples will be represented by: varicose veins (for varicectomies), carotid/femoral plaque (for thromboendarterectomy), artery wall (for aneurysmectomy/limb amputations). Alongside the collection of these samples, 5 ml of venous blood will also be collected from a peripheral venous access already positioned on the patient for the surgical procedure, regardless of the study in question.

The study requires that the samples taken be temporarily stored in order to guarantee correct analysis, according to the methods described below, and destroyed at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (age > 18 years)
* consent to participate in the study,
* patients coming to the Vascular Surgery Unit I of the IRCCS Policlinico San Donato for a vascular pathology of the arterial or venous district worthy of surgical treatment.

Exclusion Criteria:

* minor patients,
* patients who have not given their consent to participate in the study,
* patients who have vascular pathologies of the arterial or venous district not susceptible to surgical intervention.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients coming to the Operative Unit of Vascular Surgery at IRCCS Policlinico San Donato, needing open surgical intervention for arterial and/or venous pathologies
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2023-09-28 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
T-Mem expression | through study completion, an average of 2 years
  Analysis of the gene expression profile in different vascular and blood samples.

SECONDARY OUTCOMES:
3D organoids | through study completion, an average of 2 years
  Generation of pathological 3D organoids from patient vascular samples, to study the modulation of gene expression, also using sequencing techniques.

CONTACTS AND LOCATIONS:
Locations (1):
- I.R.C.C.S. Policlinico San Donato, San Donato Milanese, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Virani SS, Alonso A, Benjamin EJ, Bittencourt MS, Callaway CW, Carson AP, Chamberlain AM, Chang AR, Cheng S, Delling FN, Djousse L, Elkind MSV, Ferguson JF, Fornage M, Khan SS, Kissela BM, Knutson KL, Kwan TW, Lackland DT, Lewis TT, Lichtman JH, Longenecker CT, Loop MS, Lutsey PL, Martin SS, Matsushita K, Moran AE, Mussolino ME, Perak AM, Rosamond WD, Roth GA, Sampson UKA, Satou GM, Schroeder EB, Shah SH, Shay CM, Spartano NL, Stokes A, Tirschwell DL, VanWagner LB, Tsao CW; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2020 Update: A Report From the American Heart Association. Circulation. 2020 Mar 3;141(9):e139-e596. doi: 10.1161/CIR.0000000000000757. Epub 2020 Jan 29. PMID 31992061
- [Result] Tian K, Xu Y, Sahebkar A, Xu S. CD36 in Atherosclerosis: Pathophysiological Mechanisms and Therapeutic Implications. Curr Atheroscler Rep. 2020 Aug 9;22(10):59. doi: 10.1007/s11883-020-00870-8. PMID 32772254
- [Result] Cocola C, Magnaghi V, Abeni E, Pelucchi P, Martino V, Vilardo L, Piscitelli E, Consiglio A, Grillo G, Mosca E, Gualtierotti R, Mazzaccaro D, La Sala G, Di Pietro C, Palizban M, Liuni S, DePedro G, Morara S, Nano G, Kehler J, Greve B, Noghero A, Marazziti D, Bussolino F, Bellipanni G, D'Agnano I, Gotte M, Zucchi I, Reinbold R. Transmembrane Protein TMEM230, a Target of Glioblastoma Therapy. Front Cell Neurosci. 2021 Nov 17;15:703431. doi: 10.3389/fncel.2021.703431. eCollection 2021. PMID 34867197